CLINICAL TRIAL: NCT00294450
Title: Pouching of Fistula - a Non-comparative, Multi-center Investigation
Brief Title: Feasibility Study of a New Fistula Pouching System
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DK140OS
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2012-02-01 (Estimated); Status verified 2012-01

CONDITIONS: Cutaneous Fistula
MeSH Terms: conditions — Cutaneous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Fistula Pouching System — 3 different sizes of fistula pounching system
  Other Names: Fistula and Wound Management System

SUMMARY:
The purpose of this investigation is to carry out a clinical evaluation of a newly developed fistula pouching system's ability to function as a good pouch for fistulas, with the opening on the skin of the stomach or in a wound on the skin of the stomach.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Capable of giving informed consent
* Have to be hospitalized
* Have a fistula with the opening on the skin in the abdominal area

Exclusion Criteria:

* Pregnant and/or breast-feeding
* Receiving radiation- or chemotherapy during the investigation period

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2006-02; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Nurse's preference to use the test product in the future | Up to 18 days

CONTACTS AND LOCATIONS:
Overall Officials: Thais Benjamin N. Christensen, M.Sc. (BME), Study Chair — Coloplast A/S
Locations (7):
- United States (7):
  - St. Francis Hospital and Medical Center, Hartford, Connecticut
  - Morton Plant Hospital, Clearwarter, Florida
  - Fairview Southdale Hospital, Edina, Minnesota
  - University of Minnesota Medical Center Fairview - Riverside, Minneapolis, Minnesota
  - University of Minnesota Medical Center Fairview, Minneapolis, Minnesota
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Presbyterian Hospital of Dallas, Dallas, Texas